CLINICAL TRIAL: NCT02675647
Title: Heparin Management for Cardiopulmonary Bypass in Cardiac Surgery: A Prospective, Comparative and Randomized Study Evaluating a Dosage Based on the Ideal Body Weight in Obese Patients
Brief Title: Heparin Based on Ideal Body Weight for Cardiopulmonary Bypass in Obese Patients
Acronym: HEPOIRINE
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 6124
Record Dates: First submitted 2015-11-26; First posted 2016-02-05 (Estimated); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Surgery; Cardiopulmonary Bypass; Obese Patients (BMI ≥ 30 kg/m²)
MeSH Terms: interventions — Heparin; Cardiopulmonary Bypass

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention group (Experimental): Obese patients, randomized to receive an initial IV bolus of Heparin, before beginning of the cardiopulmonary bypass, at the dosage of 340 UI/kg based on ideal body weight of the obese patients.
  The objective is to obtain an ACT target ≥ 400 s before the beginning of CPB. If necessary, additional boluses of heparin are administered at the dose of 100 UI/kg based on ideal body weight, to maintain this target during the CPB.
  Interventions: Drug: Heparin, IV route, based on patients body weights (UI/kg); Procedure: Cardiopulmonary bypass; Drug: Protamin administration
- Control group (Active Comparator): Obese patients, randomized to receive an initial IV bolus of Heparin, before beginning of the cardiopulmonary bypass, at the usual dosage of 300 UI/kg based on total body weight of the obese patients.
  The objective is to obtain an ACT target ≥ 400 s before the beginning of CPB. If necessary, additional boluses of heparin are administered at the dose of 100 UI/kg based on total body weight, to maintain this target during the CPB.
  Interventions: Drug: Heparin, IV route, based on patients body weights (UI/kg); Procedure: Cardiopulmonary bypass; Drug: Protamin administration

INTERVENTIONS:
Drug: Heparin, IV route, based on patients body weights (UI/kg)
Procedure: Cardiopulmonary bypass
Drug: Protamin administration

SUMMARY:
The optimal heparin regimen during cardiopulmonary bypass (CPB) has not been well established in obese patients.

Results of a preview study show that the standard heparin management based on total body weight in obese patients during CPB resulted in excessive heparin level, which could lead to excessive postoperative bleeding.

To avoid this overdosing, an initial heparin bolus based on ideal body weight in obese patients was proposed.

The main objective of the study is to evaluate the effects of heparin injection, based on ideal body weight, on intraoperative plasma heparin levels and activated coagulation time (ACT) in a population of obese patients, compared to a group of obese patients undergoing CPB surgery with heparin management based of total body weight.

The secondary objectives are to evaluate the relationship between heparin level and ACT in each group of patients and at different time points during CPB, and to compare the incidence of bleeding, intraoperative transfusions and complications in the two groups of patients.

ELIGIBILITY:
Inclusion criteria:

* Obese patients (BMI ≥ 30 kg/m²)
* Planned cardiac surgery under cardiopulmonary bypass
* Coronary-artery bypass graft, or valve surgery)
* Age ≥ 18 yo

Exclusion criteria:

* Allergy to heparin
* Emergency surgical intervention
* Redo surgery
* Heart transplantation
* Surgery for circulatory assistance
* Pre-operative heparin use

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-12 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Plasma heparin level (anti-Xa activity, in UI/ml) | at 3 minutes after the first heparin injection

SECONDARY OUTCOMES:
Activated Clotting Time | during the intervention
Plasma Antithrombin III level | during the intervention at 3 minutes after heparin injection (=T1)
numbers of labile blood products transfused | during the surgery and the first 24 hours in ICU
Postoperative bleedings | during the first 24 hours in ICU, based on chest tube outputs

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpitaux Universitaires de Strasbourg, Strasbourg, France

REFERENCES:
- [Result] Vienne M, Haas E, Wipf T, Grunebaum L, Levy F, Sattler L, Hoang Minh T, Severac F, Tacquard C, Collange O, Mertes PM, Steib A. Adjusted calculation model of heparin management during cardiopulmonary bypass in obese patients: A randomised controlled trial. Eur J Anaesthesiol. 2018 Aug;35(8):613-620. doi: 10.1097/EJA.0000000000000784. PMID 29521662